CLINICAL TRIAL: NCT07190547
Title: The Effect of the Helfer Technique and ShotBlocker Application on Pain, Fear, and Anxiety in Children Receiving Intramuscular Injections: A Randomized Controlled Trial
Brief Title: Helfer Technique and ShotBlocker in Reducing Pain, Fear, and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nalan Yalçınkaya Sezer
Record Dates: First submitted 2025-07-18; First posted 2025-09-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Children; Preschool; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (ShotBloker ) (Experimental): ShotBloker
  Interventions: Other: ShotBloker
- Control group (No Intervention)
- intervention group (helper skin tap) (Experimental)
  Interventions: Other: Helfer skin tap

INTERVENTIONS:
Other: ShotBloker — ShotBlocker is a flat, horseshoe-shaped device used to reduce pain during subcutaneous or intramuscular (IM) injections. It features short, blunt, non-sharp projections approximately 2 mm in height and is designed to be placed against the skin, with a central opening that exposes the injection site. The device is applied to the skin just prior to injection, with its textured surface making contact with the skin. Although the projections do not penetrate the skin, they are believed to create a sensory stimulus associated with pain modulation based on the gate control theory.
  Arms: intervention group (ShotBloker )
Other: Helfer skin tap — Helfer Skin Tap Technique:
  After determining the injection site, gently tap the skin several times with the fingertips of the dominant (most commonly used) hand for approximately 5 seconds to relax the muscle. After the skin is wiped with antiseptic solution and stretched, the cap of the syringe in the dominant (most commonly used) hand is opened. A large V is made with the thumb and index finger of the non-dominant hand. The skin is tapped three times quickly using the whole hand to stimulate the major muscle fibers. The nurse/midwife counts to 3, and the needle is inserted into the muscle at a 90-degree angle simultaneously. To remove the needle from the skin, the skin is tapped three times quickly (again in a V shape) with the whole non-dominant hand, and the needle is withdrawn simultaneously with the final tap (tapping).
  Arms: intervention group (helper skin tap)

SUMMARY:
Various methods can be used to reduce pain experienced by children in emergency departments. However, the most critical requirement is that the method used must provide fast and effective results. Accordingly, it is essential that interventions in emergency settings are performed in a way that minimizes pain and anxiety in children and helps prevent the long-term consequences of pain (1, 2). Recently, the Helfer Skin Tap Technique (HSTT)-used to reduce stress and pain-and the ShotBlocker®, a device with small projections designed to reduce pain when applied to the skin, have gained attention (3,4,5). ShotBlocker is a non-invasive, U-shaped plastic device with small bumps, used to decrease injection-related pain, especially in children who are highly sensitive to pain (6).

In addition, a device known as Buzzy®, shaped like a bee and combining external cold application with vibration, is also commonly used. It has been proven effective in reducing pain during invasive procedures such as intramuscular (IM) injections and IV line insertions in pediatric patients (7,8). The analgesic effect of the Buzzy® device is attributed to two main mechanisms: reduced signal transmission in peripheral nerves and the gate control theory. The application of cold and vibrational stimuli to the skin activates tactile receptors, leading to the release of endogenous opioids and a subsequent decrease in pain perception (8).

Reducing pain and fear during IM injections-one of the most common painful procedures in pediatric emergency departments-is a key midwifery/nursing intervention. The authority of midwives and nurses to use non-pharmacological methods during IM injections is clearly defined in their respective professional regulations. Given the nature of pediatric emergency units, midwives and nurses contribute significantly to increasing both child and parent comfort by using practical, fast-acting, and low-cost methods that can be easily implemented during painful procedures.

Demonstrating the positive effects of non-pharmacological methods on reducing pain and fear in children of different age groups during IM injections is crucial, both for enriching the literature and for encouraging the widespread use of evidence-based, cost-effective practices in clinical settings. Making such approaches a routine part of care delivery in pediatric units is of great importance.

The aim of the study was to investigate the effects of ShotBlocker and HSTT on the pain and fear experienced by children aged 4-6 years during IM injection in pediatric emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 6 years,
* An intramuscular (IM) medication order was prescribed by a physician,
* The IM injection was administered in the pediatric emergency department,
* No history of chronic pain-causing illness,
* No diagnosis of neurodevelopmental disorders,
* Had not received any analgesic medications in the past 6 hours,
* No history of syncope (fainting) during previous injections,

No diagnosis of mental retardation,

* No scar tissue or muscle atrophy at the intended injection site,
* Body mass index (BMI) percentile between the 10th and 90th percentiles for age and gender,
* Both child and parent provided informed consent to participate in the study.

Exclusion Criteria;

* Participants were excluded from the study if:
* The child was younger than 4 or older than 6 years,
* There was scar tissue or muscle atrophy at the injection site,
* The child or parent had communication difficulties,
* The child's BMI was below the 10th percentile (cachectic) or above the 90th percentile (obese),
* Either the child or parent declined to participate in the research.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Measurement Tool | 12 weeks
  he Wong-Baker FACES Pain Rating Scale was used to assess self-reported pain levels. This scale consists of six facial expressions ranging from "no hurt" (0) to "hurts worst" (10), allowing children to select the face that best represents their level of pain.
Assessment Time | 12 weeks
  Pain scores were recorded immediately after the injection.Developed by Wong and Baker, it features six hand-drawn facial expressions on a horizontal plane. Scored from 0 to 10, the leftmost face features a smiling face, representing "no pain." Pain increases from left to right. The rightmost face features a face with tears, representing "unbearable pain."
Measurement Tool (Fear Level) | 12 weeks
  The Children's Fear Scale was used to assess the child's level of fear. This visual scale consists of five facial expressions depicting increasing levels of fear (scores range from 0 to 4). from neutral expression (0=no anxiety) to frightened face (4=severe anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethically, patient information can be shared upon reasonable request without revealing their identities for security reasons.